CLINICAL TRIAL: NCT01020240
Title: Effectiveness of an Orientation Guide for Puerperal Women After Cesarean.
Brief Title: Physiotherapy in Postpartum After a Cesarean
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sao Marcos University (Other)
Responsible Party: Patricia Andrade Batista, São Marcos University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Unimarco
Record Dates: First submitted 2009-11-24; First posted 2009-11-25 (Estimated); Last update posted 2009-11-26 (Estimated); Status verified 2009-11

CONDITIONS: Postpartum Period
Keywords: Immediate puerperium; physiotherapy in postpartum; cesarean complications

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Avaliation (No Intervention): This group will have 15 women in puerperium and will be realize an interview to avalide the cesarean discomforts in immediate puerperium. These dates will be use for elaborate the orientations guide.
  Interventions: Behavioral: Avolition
- Orientation (No Intervention): In this group will be realize an interview to avalide the cesarean discomforts in immediate puerperium or in the first post operatory and in the second post operatory wil be realize a new interview.
  Interventions: Behavioral: Orientation
- Guide (Experimental): in This group wiil be realize an interview to avalide the cesarean discomforts in immediate puerperium or in the first post operatory, will be realize the orientations and the guide will be give, and in the second post operatory will be realize a new interview.
  Interventions: Behavioral: Guide

INTERVENTIONS:
Behavioral: Avolition — - avolition for cesarean discomforts
  Arms: Avaliation
Behavioral: Orientation — * avolition of cesarean discomfort
  * physiotherapy orientation
  Arms: Orientation
Behavioral: Guide — * avolition of cesarean discomfort
  * physiotherapy orientation
  * guide orientation
  Arms: Guide

SUMMARY:
The purpose of this study is to promote a prevention of the complications using an elaborate guide effective and easy to understand.

DETAILED DESCRIPTION:
The puerperium consists the period of pregnancy and postpartum cycle that the alterations provoked for pregnancy and delivery on the women organism return to your state before pregnancy. The physiotherapist can follow the puerperium since hospital phase until women has been recovered of pregnancy physiologist alterations.

ELIGIBILITY:
Inclusion Criteria:

* have between 15 and 35 yeas old
* has realize an emergency or elective cesarean
* being in immediate puerperium and did not have receive any orientation

Exclusion Criteria:

* complications in delivery and postpartum
* complications with the baby
* physicologics disease

Ages: 15 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45 (Actual)
Dates: Start 2009-03; Primary Completion 2009-05 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Analogic Visual Scale | 6 months

SECONDARY OUTCOMES:
Analogic Visual Scale | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Batista, Principal Investigator — São Marcos University
Locations (1):
- Sepaco Hospital, São Paulo, São Paulo, Brazil